CLINICAL TRIAL: NCT06796335
Title: Development and Implementation of an Intervention Enhancing Involvement of Relatives to Patients With Acquired Brain Injury or Malignant Brain Tumour
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Hvidovre University Hospital (Other); Regionshospitalet Hammel Neurocenter (Other)
Responsible Party: Principal Investigator, Rikke Guldager, Head of Nursing Research, Rigshospitalet, Denmark
Other Study IDs: ID P-2022-733
Record Dates: First submitted 2025-01-20; First posted 2025-01-28 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Brain Injury; Brain Tumor Adult; Traumatic Brain Injury; Glioblastoma
Keywords: Involvement; Relatives; Complex intervention; Qualitative research; nurse intervention; tool; dialog
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic; Glioblastoma; Margins of Excision

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ABI (Aquired Brain Injury)
  Interventions: Other: RIGht
- ABI (Aquired Brain Injury), MBT (Malignant Brain Tumor): The study will be conducted in six inpatient units in two hospice sites in Denmark that admitted adult patients with respectively acquired brain injury and malignant brain tumor.
  Interventions: Other: RIGht

INTERVENTIONS:
Other: RIGht — The final intervention consists of five components; 1) education of nurses 2) a dialog tool used in a single session intervention and follow- up 3) a relative- to- relative list 4) video material 5) guidelines on how to document the relative involving plan in the patient's electronic journal.

SUMMARY:
Caring for a loved one with a serious illness like acquired brain injury (ABI) or primary malignant brain tumors (PMBT) can be a challenging and burdensome experience, often affecting the well-being and quality of life of relatives. While family and friends can provide some support, this is not always enough to address the diverse needs of caregivers. Relatives often have different requirements for support, information, and involvement in the patient's care. Understanding these varying needs is key to ensuring both the patient and their caregivers are effectively supported during the illness journey.

This study aims to develop and test an intervention that helps healthcare professionals better support relatives in their caregiving role. The intervention uses a dialogue tool, which is designed to help nurses assess and follow up on the differing needs of relatives for involvement in the care of patients with ABI and PMBT. The goal is to enhance the experience of both the patient and their caregivers throughout the illness process.

The study will take place across seven units in two regions of Denmark, and it involves relatives of patients with ABI or PMBT. The main questions the study aims to answer are:

* Can an intervention that involves relatives improve their role in the care of patients with ABI and PMBT?
* Will this intervention help both patients and their relatives feel more supported and satisfied during the treatment process?

Participants will receive support through an intervention that includes several key components:

* Nurse training on how to use the dialogue tool to assess and address the varying needs of relatives for involvement.
* A list created by relatives, for relatives, to share experiences and advice with one another.
* Video materials explaining the background and purpose of the intervention to help relatives understand how it can benefit them.
* Guidelines for documenting the involvement of relatives in the patient's electronic health record.

By offering targeted support to relatives, this intervention aims to enhance their involvement in the treatment process, ensuring that both patients with ABI or PMBT and their families are better supported throughout the course of the illness.

DETAILED DESCRIPTION:
Background Relatives of patients with acquired brain injury (ABI) or primary malignant brain cancer (WHO grade III and IV) often face substantial caregiving burdens, which increase the risk of anxiety and depression. The patient's condition can significantly alter the daily lives of relatives, many of whom assume long-term caregiving responsibilities. These challenges are compounded by the emotional and practical difficulties faced by families, particularly when patients experience significant cognitive, physical, and emotional impairments. In cases of ABI, relatives often witness a gradual or sudden decline in the patient's functioning, leading to a profound sense of loss and a shift in family roles. Similarly, relatives of patients with PMBT are faced with the rapid progression of the disease, which demands constant adjustment to their caregiving responsibilities.

Despite these challenges, research underscores the importance of involving relatives in the patient's care and treatment, as this involvement has been shown to improve patient outcomes and family satisfaction. Furthermore, it promotes better communication and collaboration between healthcare professionals and families, which is essential for the rehabilitation process. However, Denmark currently lacks a validated tool to assess the diverse needs of relatives during treatment and rehabilitation, considering their individual resources and capacities. This gap leaves healthcare professionals without a standardized means to engage relatives in a way that is both meaningful and beneficial for the patient's recovery.

Furthermore, no intervention studies have specifically targeted the active engagement of relatives of patients with ABI or PMBT to provide direct support to relatives and indirectly benefit the patient. Given the growing body of evidence that highlights the importance of tailored support for relatives, there is an urgent need for a structured and evidence-based approach that can address the varying needs of families in different clinical settings.

Purpose The primary aim of this study is to develop, pilot, and evaluate a tool designed to identify and address the varied needs and resources of relatives. This tool will ensure that the involvement needs of relatives are assessed throughout the patient's treatment and rehabilitation. Specifically, the tool will help identify the unique challenges faced by relatives based on their socio-economic, emotional, and practical circumstances, thereby providing a personalized support framework. This systematic approach aims to reduce caregiver strain, improve the well-being of relatives, and enhance the overall rehabilitation process for the patient.

Methods The intervention was developed using the Medical Research Council's framework for complex interventions, with a focus on the participation of both relatives and healthcare professionals. The development process was iterative, incorporating theoretical models, evidence-based practices, and practical insights from caregiving contexts. Data was gathered through scoping reviews, field observations, and discussions with relatives and nurses across seven healthcare units in two regions of Denmark. These discussions provided diverse perspectives on the challenges faced by relatives in different clinical settings, including the specific needs of families coping with ABI and glioblastoma.

Through this process, it became evident that relatives experience a wide range of needs, from emotional and psychological support to practical assistance with caregiving tasks. This input directly influenced the design of the intervention, ensuring that it would be both comprehensive and responsive to the varying circumstances of families.

Results

The intervention consists of five key components:

1. Nurse education: Equipping healthcare professionals to better support and involve relatives in the patient's care.
2. A dialogue tool: For structured conversations between healthcare professionals and relatives to address specific needs.
3. A relative-to-relative list: Tips for navigating the healthcare system, including guidance on how to access available resources, such as financial support, social services, and patient advocacy groups, which can help alleviate the strain on families.
4. Video resources for caregivers: A video explaining the background and rationale for the intervention, featuring stories from relatives sharing their experiences.
5. Guidelines for documenting relative involvement in the patient's electronic health record: Standardized tracking of relative participation in care.

A panel of 18 relatives, selected based on geographic location, age, and gender, contributed to the development and evaluation of the intervention. Their roles ranged from informants to advisors, providing feedback on activities, refining ideas, and assisting in the creation of materials, such as videos and the relative-to-relative list. Additionally, they played a crucial role in training nurses, ensuring that the intervention met the needs of families in a real-world healthcare context.

Clinical Perspectives The standardized tool is expected to systematically assess the needs and resources of relatives, ensuring tailored support according to their circumstances. By recognizing that relatives of patients with ABI and PMBT have different needs based on their personal situation and available resources, the tool aims to offer a more personalized and effective intervention. This personalized approach is anticipated to improve relative satisfaction, enhance their sense of agency in the caregiving role, and contribute to the rehabilitation process for the patient.

The intervention also aims to improve communication and collaboration between relatives and healthcare professionals. By fostering a more supportive environment for both patients and families, the intervention is expected to lead to better care outcomes, greater family satisfaction, and a more efficient healthcare process. Ultimately, this will contribute to an overall improvement in the patient's rehabilitation and long-term quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Relatives of adult patients with an acquired brain injury or primary malignant brain tumor
* Patients most be hospitalized
* Patients must agree to give their informed consent to involve their relatives
* Able to read and understand english

Exclusion Criteria:

* Relatives under the age of 18 years of age

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is conducted in six inpatient units in two hospice sites in Denmark that admitted adult patients with respectively acquired brain injury and malignant brain tumor. Acquired brain injuries often occur suddenly and unexpectedly. Suffering from an acquired brain injury has major consequences, not only for the patients, due to the devastating impact on their physical, cognitive, social, and psychological well-being, but also for the relatives who may need to take on a lifelong role as carers
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Focus group interviews | Op til 6 weeks post intervention
  Themes describing nurses evaluation of the acceptability and fidelity of the intervention will be evaluated i through qualitative focus group interviews. A Thematic analysis as suggested by Braun and Clark will be conducted.

SECONDARY OUTCOMES:
PEIRS-22 | Op til 6 weeks post intervention
  To evaluate the relatives' experience of being involved in the research process, the Patient Engagement in Research Scale (PEIRS-22) is being utilized. This tool measures the degree of meaningful participation on a scale from 0 to 100, where a high score reflects a high level of meaningful engagement in the research.
Semi-structured interviews | Op til 10 weeks post intervention
  To evaluate the acceptability, relevance, and apprropriateness semi-structured interviews will be conducted with relatives who received the intervention. Data will be analysed utilizing Braun and Clarks' thematic analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Department of neurosurgery, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Not relevant for this study

REFERENCES:
- [Background] Guldager R, Nordentoft S, Poulsen I, Aadal L, Loft MI. Wants and needs for involvement reported by relatives of patients with a malignant brain tumor: a scoping review. JBI Evid Synth. 2023 Nov 1;21(11):2188-2210. doi: 10.11124/JBIES-22-00311. PMID 37435678
- [Background] Lundh MG, Nordentoft S, Smedegaard PS, Aadal L, Loft MI, Poulsen I, Guldager R. Interventions facilitating the involvement of relatives of patients with acquired brain injury or malignant brain tumour: A scoping review. J Clin Nurs. 2025 Mar;34(3):784-794. doi: 10.1111/jocn.17328. Epub 2024 Jul 30. PMID 39078079
- [Background] Guldager R, Nordentoft S, Aadal L, Loft MI, Poulsen I. Wants and needs of relatives' involvement in patient care: the same but different. JBI Evid Synth. 2023 Nov 1;21(11):2154-2155. doi: 10.11124/JBIES-23-00469. No abstract available. PMID 37935421
- [Background] Guldager R, Nordentoft S, Poulsen I, Aadal L, Loft MI. Wants and needs for involvement experienced by relatives of patients with an acquired brain injury: a scoping review. JBI Evid Synth. 2023 May 1;21(5):886-912. doi: 10.11124/JBIES-22-00022. PMID 36729839